CLINICAL TRIAL: NCT00822003
Title: Effects of Oral GLP-1 on Glucose Homeostasis and Appetite Profile Following an Oral Glucose Tolerance Test in Healthy Male Subjects
Brief Title: Effects of Oral GLP-1 on Glucose Homeostasis and Appetite Profile in Healthy Male Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Beglinger Christoph, Prof. Dr.med., University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EKBB 127/07, Amendment 1
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Glucose Homeostasis
Keywords: GLP-1; insulin; glucose
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Human GLP-1
  Interventions: Drug: Oral GLP-1
- 2 (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral GLP-1 — GLP-1 tablet (2mg)
  Arms: 1
Drug: Placebo — Control tablet
  Arms: 2

SUMMARY:
The investigators aimed to investigate the pharmacokinetic and pharmacodynamic effects of a single dose (2 mg) of oral GLP-1 administered prior to an oral glucose tolerance test (oGTT) in 16 healthy males

DETAILED DESCRIPTION:
Background: Glucagon like peptide-1 (GLP-1) promotes satiety and reduces food intake. GLP-1 is secreted from intestinal L-cells into the splanchnic circulation, it is (i) subject to rapid breakdown and (ii) submitted to a high liver extraction. Highest concentrations of GLP-1 are therefore found in the splanchnic blood rather than in the systemic circulation. An oral delivery system would mimick the physiological path of endogenous secretion. Objective: We aimed to investigate the pharmacokinetic and pharmacodynamic effects of a single dose (2 mg) of oral GLP-1 administered prior to an oral glucose tolerance test (oGTT) in 16 healthy males.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* no gastrointestinal or endocrine disorder

Exclusion Criteria:

* females
* alcohol or drug abuse
* active virus hepatitis

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

SECONDARY OUTCOMES:
Glucagon secretion GH release adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — Clinical Research Center, University Hospital Basel
Locations (1):
- Clinical Research Center, University Hospital Basel, Basel, Canton of Basel-City, Switzerland